CLINICAL TRIAL: NCT05814536
Title: A Phase I, Multi-center, Open-label, Single-arm Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of AB-218 for Treating Adult Patients With Advanced IDH1 Mutant Cholangiocarcinoma and Other Solid Tumors
Brief Title: IDH1 Inhibitor AB-218 in Patients With Advanced IDH1 Mutant Cholangiocarcinoma and Other Solid Tumor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor adjusted the study strategy
Sponsor: AnHeart Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-218-G104
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Cholangiocarcinoma With IDH1 Mutation; Solid Tumors With IDH1 Mutation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AB-218 (Experimental): AB-218 for the treatment of adult patients with advanced cholangiocarcinoma, chondrosarcoma and other solid tumors with IDH1 mutation.
  Interventions: Drug: AB-218 capsule

INTERVENTIONS:
Drug: AB-218 capsule — Take AB-218 orally twice daily, ideally with 12 hours between doses (and a minimum of 8 hours between doses), at a dose assigned by the study. The study treatment is defined as occurring in 28-day cycles with continuous dosing. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs earlier.

SUMMARY:
This is an open label, single-arm Phase I study to evaluate the safety, tolerability, PK and preliminary efficacy of AB-218, an oral IDH1 inhibitor, for the treatment of adult patients with advanced IDH1 mutant cholangiocarcinoma and other solid tumors who have failed at least one prior therapy in the advanced stage.

The study contains a dose escalation part and a dose expansion part. In the dose escalation part, participants are enrolled sequentially into one of 3 dose levels of AB-218 (125 mg BID, 250 mg BID and 500 mg BID) following a 3+3 rule. Intensive PK sampling will be performed during the dose escalation part. Participants will be followed up for DLTs from the date of first study dose to 28 days afterwards. When all participants in the dose escalation part have completed the 28-day DLT observation period, SMC will review the available data including but not limited to safety, tolerability and PK, and then recommend the dose for the study dose expansion part.

In the dose expansion part, there are 2 disease cohorts planned: cholangiocarcinoma (CCA) and other IDH1 mutant solid tumors. It is planned to enrol 30 participants in the CCA cohort and another 15 participants in other IDH1 mutant solid tumors, to assess the safety and preliminary efficacy of AB-218. Sparse PK samples will be collected to further evaluate the PK profile in the different target populations.

Each participant will undergo screening up to 28 days prior to the start of the treatment period. The treatment period consists of a visit on Day 1 of every 28-day cycle and continues until any of disease progression, unacceptable toxicity, withdrawal of consent or death. An end of treatment (or early discontinuation) visit occurs 30 days (± 7 days) after the last dose of study medication, and a survival follow call every 12 weeks until death, withdrawal of informed consent, loss to follow-up (LTFU) or termination of the study by the sponsor, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 years of age at the time of signing the informed consent form.
2. Must have locally advanced or metastatic solid tumors that have recurred or progressed following treatment with at least 1 prior systemic therapy, or that have not responded to prior systemic therapy; or the patient is unfit for any intensive chemotherapy in the first line setting.
3. Must have histologically confirmed IDH1 mutation from testing of a primary or metastatic tumor before first study treatment. Patients must have archival primary tumor biopsy or surgical specimens, or biopsies of recurrence of metastasis for IDH1 mutation confirmation and status of other concurrent gene mutations. Patients shall provide formalin-fixed paraffin-embedded (FFPE) tissue slides without staining, which are shipped to the designated laboratory. The IDH1 mutation must be determined by a validated assay as performed in Clinical Laboratory Improvement Amendments (CLIA)-certified/College of American Pathologists (CAP)-accredited or locally equivalent clinical laboratories. Patients whose tumors have not been tested for IDH1 mutation, must be consented with the pre-screening ICF to allow collection of tumor tissue and testing at the designated qualified central laboratory. These patients may only be consented to the study with the full ICF if they have a documented IDH1 mutation.
4. Must have a measurable lesion(s) as per the RECIST v1.1 criteria.
5. Patients with chronic HCV infection are acceptable to enroll, if ≥ 4 weeks between achieving sustained viral response and start of study drug. Anti-viral therapy is allowed during the study treatment period.
6. Patients with chronic HBV infection may enroll in the study, if HBV DNA is <1000 copies/mL prior to the start of study treatment. Anti-viral therapy is allowed during the study treatment period.
7. Must have life expectancy ≥ 3 months.
8. Must have Eastern Cooperative Oncology Group (ECOG) performance status (PS) score ≤ 1.
9. Must have a Child-Pugh class A liver score within 7 days prior to first dose of study treatment.
10. Must have adequate organ functions as defined below:

    Absolute neutrophil count (ANC)≥ 1.5 X 109/L, Hemoglobin≥ 80 g/L Creatinine Clearance* (Cockcroft-Gault Formula) ≥ 60 mL/min Total Bilirubin≤ 2 x ULN,≤ 3 x ULN, for participants with documented Gilbert's syndrome AST and ALT≤ 5 x ULN, Albumin≥ 30 g/L, INR ≤ 1.5 x ULN unless patient is receiving anti-coagulant therapy, aPTT must be within the therapeutic range of intended use of anticoagulants
11. Adequate biliary drainage, with no evidence of ongoing infection (patients on maintenance antibiotics are eligible when acute sepsis has resolved)
12. Recovery to Grade 1 from any toxicities due to prior therapies, except conditions such as peripheral neuropathy, alopecia and irreversible changes associated with radiation therapy; peripheral neuropathy due to prior therapies must have recovered to ≤ Grade 2.
13. Female patients who engage in heterosexual intercourse must be of nonchildbearing potential, defined as either surgically sterile (i.e., hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), OR be postmenopausal with at least 1 year of amenorrhea, OR must agree to use a highly effective method of contraception from the beginning of Screening until at least 90 days after the last dose of study drug.

    • Acceptable highly effective methods of contraception include:
    * Combined estrogen-progestin oral hormonal contraception associated with consistent inhibition of ovulation.
    * Desogestrel based progestin only contraception associated with consistent inhibition of ovulation; this includes oral, injectable, and implantable methods
    * Intravaginal and transdermal hormone delivery methods
    * Intrauterine device (with or without hormone elution)
    * Bilateral tubal occlusion or ligation (must be documented)
    * Vasectomized partner (must be documented) or
    * Sexual abstinence (only when it is the usual and preferred lifestyle of the patient)
14. Male patients must agree to use a condom when sexually active with a female partner of childbearing potential from Screening until at least 90 days after the last dose of study drug (or be surgically sterile [i.e., vasectomy with documentation]; or remain abstinent [when this is in line with the preferred and usual lifestyle]. Male patients should also agree not to donate sperm for the duration of the study and until at least 90 days after the last dose of study drug.
15. Must be capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
16. Must be able to undergo the protocol-specified procedures, including blood tests, urinalysis.

Exclusion Criteria:

1. Patients diagnosed with IDH1 mutant glioma or acute myeloid leukemia (AML).
2. Patients with history or complication of any of the following diseases within 3 months prior to the initial dose of the investigational drug.

   * Myocardial infarction
   * Severe or unstable angina pectoris
   * Coronary or peripheral endovascular treatment
   * Heart failure
   * Cerebrovascular disorder including transient ischemic attack, stroke, central nervous system (CNS) bleeding.
3. Uncontrolled active systemic fungal, bacterial, or other infection (despite appropriate antibiotics or other treatment).
4. HIV infection as determined by an HIV antibody test.
5. Presence of Grade 3 ascites, as defined in the Guidance on the Management of Ascites and Complications in Cirrhosis 36. The patient has significant bloating, tests positive for shifting dullness, and may have abdominal distension leading to umbilical hernia; on assessment with ultrasound, the ascites occupies the entire abdominal cavity, and the middle abdomen is filled with ascites, with a depth of >10 cm.
6. Gastrointestinal diseases that may interfere with oral ingestion of the study drug or may affect absorption of the study drug.
7. Prior anticancer therapy, within the applicable periods shown below, before the start of the protocol treatment:

   * Systematic Therapy: within 3 weeks
   * Radical Surgery: within 3 weeks
   * Radiation therapy: within 12 weeks (excluding the palliative radiotherapy or radiotherapy on the non-target lesions)
   * Infusion of blood component or the recombinant human blood product, for example, RBC, Platelet, rhGSF: within 2 weeks
8. Have received prior anti-cancer therapy targeted to the IDH1 mutation.
9. Patients taking substrates of cytochrome CYP2C8, CYP2C9, and CYP3A4 with narrow therapeutic window, should be excluded unless they can be transferred to other medications prior to enrolling. Patients taking sensitive CYP 2C8, 2C9 or 3A4 substrate medications may require dosage adjustment unless they can be transferred to other medications within ≥ 5 half-lives prior to dosing.
10. Patients taking sensitive substrates of P-gp and BCRP transporters should be excluded unless they can be transferred to other medications prior to enrolling. Patients taking sensitive substrates of P-gp and BCRP may require dosage adjustment unless they can be transferred to other medications within ≥ 5 half-lives prior to dosing.
11. Known hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any other excipient present in the pharmaceutical form of the investigational medicinal product(s).
12. Advanced arrhythmia of Grade ≥ 2 per Common Terminology Criteria for Adverse Events (CTCAE) v5.0, uncontrolled atrial fibrillation (any grade) and QTcF >470 msec for females or >450 msec for males.
13. Pregnant or breastfeeding female patient.
14. Psychiatric disease or symptoms that may interfere with continuous participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-05-06 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
TEAEs | About 24 months
  Treatment-Emergent Adverse Events (TEAEs) including events reported following physical examination, vital signs assessment, clinical laboratory assessment or electrocardiogram (ECG)
DLT incidence | Dose escalation part, about 6 months
  Dose limiting toxicity incidence

SECONDARY OUTCOMES:
Overall Response Rate | About 24 months
  Proportion of subjects with the best overall confirmed response of complete response (CR) or partial response (PR) according to RECIST v1.1
Duration of Response | About 24 months
  Defined as the time from the first date of objective response (CR or PR) to the first documented date of disease progression. Response assessments are per RECIST v1.1 criteria and are investigator designated
Disease Control Rate | About 24 months
  Defined as the proportion of subjects with a best overall response of CR, PR or stable disease per RECIST v1.1 criteria) as assessed by the investigator
Progress Free Survival | About 24 months
  Defined as the time from first dose of AB 218 until the date of disease progression, or death from any cause. Response assessments are per RECIST v1.1 criteria and are investigator designated.
Overall Survival | About 48 months
  Defined as the time from the first dose of AB 218 to death due to any cause.
Cmax | 8 Days. At the Day1 and Day8 of Cycle1 for dose escalation part and dose expansion part(each cycle is 28 days)
  Plasma drug peak concentration
Tmax | 8 Days. At the Day1 and Day8 of Cycle1 for dose escalation part and dose expansion part(each cycle is 28 days)
  Time to reach plasma drug peak concentration
AUC8h | 8 Days. At the Day1 and Day8 of Cycle1 for dose escalation part(each cycle is 28 days)
  Area under the plasma drug concentration time curve from 0 to 8h
AUC12h | 8 Days. At the Day1 and Day8 of Cycle1 for dose escalation part(each cycle is 28 days)
  Area under the plasma drug concentration time curve from 0 to 12h
AUC6h | 8 Days. At the Day1 and Day8 of Cycle1 for dose expansion part(each cycle is 28 days)
  Area under the plasma drug concentration time curve from 0 to 6h
Ctrough | 4 Months. At the end of Cycle 4 (each cycle is 28 days).
  Trough concentration
Plasma concentration of 2-HG | 4 Months. At the end of Cycle 4 (each cycle is 28 days).
  Plasma concentration of 2-HG

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The fourth hospital of Hebei medical university, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - The Third Affiliated Hospital of the PLA naval medical university, Shanghai, Shanghai Municipality
  - Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang
  - Jinan Central Hospital, Jinan, Zhejiang